CLINICAL TRIAL: NCT04091698
Title: 11 El-Saraya St. - Manial - Cairo
Brief Title: Clinical and Biochemical Assessment of the Effect of Topical Use of Coenzyme Q10 Versus Topical Corticosteroid in Management of Symptomatic Oral Lichen Planus: Randomized Controlled Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Abdelsamie Bakry Nafie, demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Q10 in oral lichen planus
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Oral Lichen Planus
Keywords: co enzymeQ10 - Antioxidant- Corticosteroids
MeSH Terms: conditions — Lichen Planus, Oral | interventions — ubiquinol

STUDY DESIGN:
Intervention Model Description: two parallel group one take Q10 mucoadhesive tablets and other take topical corticosteroid for 3 months follow up measuring pain ,clinical size of lesion and salivary level of Malondialdehyde as oxidative biomarker
Who Masked: Outcomes Assessor
Masking Description: Double-blinded trial, outcome assessors and statistician
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical Q10 mucoadhesive tablets (Active Comparator): will receive topical co enzyme q10 in the form of mucoadhesive tablets 3 times daily for 3months.
  Interventions: Drug: Co-Enzyme Q10 mucoadhesive tablets
- topical corticosteroid (Placebo Comparator): will receive topical corticosteroid (kenacort A Orabase: triamcinolone acetonide 0.1%5gram adhesive paste - dermapharm), 4 times daily for 3months.
  Interventions: Drug: Co-Enzyme Q10 mucoadhesive tablets

INTERVENTIONS:
Drug: Co-Enzyme Q10 mucoadhesive tablets — will receive topical co enzyme q10 in the form of mucoadhesive tablets 3 times daily for 3months.
  Other Names: Q10 mucoadhesive tablets -ubiquinol

SUMMARY:
The aim of the present investigation is to assess the clinical therapeutic effect of topical use of Coenzyme Q10 versus topical corticosteroid in management of symptomatic oral lichen planus and determine whether the effect, if any, was due to its antioxidant activity.

DETAILED DESCRIPTION:
Oral lichen planus (OLP) is a relatively common chronic inflammatory mucocutaneous autoimmune disease that primarily affects the skin and mucosal surfaces including the oral cavity with a variety of clinical manifestations including reticular, papular, hyperkeratotic, atrophic, erosive, and bullous forms 1,2. The erosive, atrophic, and bullous type lesions are usually accompanied with pain or burning sensation that affects the patient's quality of life3. Intraorally, the buccal mucosa, dorsum of the tongue and the gingiva are commonly affected 4 .OLP has most often been reported in middle aged patients3. Women account for 60% to 75% of patients with OLP 5.

OLP is estimated to affect1% to 2.0% of the general population. Around 40% of lesions occur on both oral and cutaneous surfaces, 35% occurs on cutaneous surfaces alone, and 25% occur on oral mucosa alone 6,7.

Several predisposing factors might be involved in the pathogenesis of OLP. Earlier studies have implicated stress, anxiety and depression as possible factors. Familial cases of OLP have been reported and the role of genetic predisposition was considered8.

The exact etiology of OLP is still unknown, but cell-mediated immune dysfunction is implicated in the complex etio-pathogenesis of this disease. Large amounts of cytokines that are released by affected keratinocytes and the associated inflammatory elements play a key role in the selective recruitment of cytotoxic CD8+ T cells trigger apoptosis of the basal cells of the oral epithelium. T-cell dominated infiltrate in the sub epithelial region, which characterizes OLP, induces further release of cytokines9.

Cytokines may be produced by nearly every cell, but mostly act locally on cell receptors and have high potency10. Their production gives rise to an inflammatory cascade. One of the most important elements in this cascade is overexpression of tumor necrosis factor-alpha (TNF- α). TNF- α causes tissue destruction and overproduction of other cytokines, especially interleukin (IL)-6 which, in turn, leads to further inflammation and tissue degradation 11. Production of cytokines can in turn stimulate production of Reactive Oxygen Species (ROS) and cause oxidative damage to the tissues 12 .

Malondialdehyde (MDA), as the lipid peroxidation marker, increases in an oxidative stress-dependent situation 13. Actually, higher levels of MDA were reported in serum and saliva of patients affected by OLP14-17.

A variety of treatments have been proposed for OLP: topical or systemic corticosteroids, cyclosporine, retinoids, azathioprine, tacrolimus, pimecrolimus, photo chemotherapy, and surgery 18.

Systemic and topical corticosteroids are probably the most effective treatment modality for patients with diffuse erosive OLP or multisite disease 19 .Despite the therapeutic effects of corticosteroids, they have significant morbidity and disturbing adverse effects such as fungal infections and adrenal suppression. Moreover, steroid use is contraindicated in patients who are breastfeeding, and have to be used with caution in patients with herpetic infections, glaucoma, HIV infection, tuberculosis, diabetes mellitus, candidiasis, and hypertension, as well as in pregnant women, resulting in a continuing search for novel therapies 20.

Coenzyme Q10 (CoQ10) or ubiquinone is a lipid-soluble vitamin-like antioxidant naturally found in the diet and can also be synthesized endogenously by all cells of our body. It is one of the key components in ATP production in ETC. CoQ10 protects membranes against oxidation, and regenerates vitamins E and C and enzymatic antioxidant systems, and modulates prostaglandin metabolism 21, 22.

The maximal antioxidative power of the CoQ10 coenzyme is credited to its electron-donating properties that neutralize free radicals 23, and its ability to replenish other valuable endogenous antioxidants 24.

CoQ10 is located in the membranes in close proximity to the unsaturated lipid chains to act as a primary scavenger of free radicals and prevent lipid peroxidation 25.. Any certain condition that leads to increased levels of ROS (either by overproduction or impaired removal) or reduced function of antioxidants is called "oxidative stress". ROS may be toxic to cells via inactive enzymes, denaturizing proteins, DNA destruction, and lipid peroxidation. These events lead to damaged cell membrane, increased reactive aldehyde materials, and impaired cell function. The level of ROS and lipid peroxidation may be related to OLP 26,27. This suggests that oxidative stress is a major trigger for OLP, and the level of antioxidants is a potential determinant of susceptibility to be affected by OLP 28, 29.

In addition, studies have shown that CoQ10 also exerts anti-inflammatory properties via IL-1, TNF-α, and NFκB1-dependent gene expression, thus enhancing clearance of inflammation within the lesion to promote tissue regeneration and wound healing30.

Papucci et al. 31 demonstrated that treatment with CoQ10 lowered the number of apoptotic keratocytes in response to excimer laser irradiation to a much higher extent than other free radical scavengers. Moreover, supplemental CoQ10 has good safety record; no adverse effects have been reported with daily dosage ranging from 600 to 1200mg

ELIGIBILITY:
Inclusion Criteria:

1. Patients free from any systemic disease according to the detailed questionnaire of the modified Cornell Medical Index 34.
2. Patients not receiving any medication either topical or systemic that could cause lichenoid reaction during the 3 months before the study.
3. Patients diagnosed by a dermatologist and oral medicine specialist as suffering from OLP.
4. Patients clinically and histopathologically diagnosed as suffering from OLP according to World Health Organization's (WHO's) clinic-pathological diagnostic criteria for LP35.
5. Patients who agree for the biopsy in undiagnosed cases.
6. Patients who are willing to participate in this study (will give informed consent) and have the ability to complete the study.

   * Exclusion criteria:

(1) Patients taking systemic drugs such as systemic steroid, other immunosuppressive therapy for at least 8 weeks prior to the study.

(2) Patients treated with any oral topical medications for at least four weeks prior to the study.

(3) Patients with suspected restoration-related reaction. (4) Pregnant and lactating mothers.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
pain score | 3months
  visual analogue scale scoring system
clinical size of lesion | 3months
  Thongprasom score system

SECONDARY OUTCOMES:
Salivary level of Malondialdehyde | 3months
  detect by ELISA

REFERENCES:
- [Background] Scrobota I, Mocan T, Catoi C, Bolfa P, Muresan A, Baciut G. Histopathological aspects and local implications of oxidative stress in patients with oral lichen planus. Rom J Morphol Embryol. 2011;52(4):1305-9. PMID 22203938
- [Background] Sugerman PB, Savage NW, Zhou X, Walsh LJ, Bigby M. Oral lichen planus. Clin Dermatol. 2000 Sep-Oct;18(5):533-9. doi: 10.1016/s0738-081x(00)00142-5. No abstract available. PMID 11134848
- [Background] Ismail SB, Kumar SK, Zain RB. Oral lichen planus and lichenoid reactions: etiopathogenesis, diagnosis, management and malignant transformation. J Oral Sci. 2007 Jun;49(2):89-106. doi: 10.2334/josnusd.49.89. PMID 17634721
- [Background] Bhagavan HN, Chopra RK. Plasma coenzyme Q10 response to oral ingestion of coenzyme Q10 formulations. Mitochondrion. 2007 Jun;7 Suppl:S78-88. doi: 10.1016/j.mito.2007.03.003. Epub 2007 Mar 27. PMID 17482886
- [Background] Yang LL, Liu XQ, Liu W, Cheng B, Li MT. Comparative analysis of whole saliva proteomes for the screening of biomarkers for oral lichen planus. Inflamm Res. 2006 Oct;55(10):405-7. doi: 10.1007/s00011-006-5145-8. PMID 16850138
- [Derived] Abdelsamie M, Zahran F, Hussine AA, Shaker O, Al-Mahallawi AM. Clinical and biochemical assessment of the effect of topical use of coenzyme Q10 versus topical corticosteroid in management of symptomatic oral lichen planus: randomized controlled clinical trial. BMC Oral Health. 2023 Jul 21;23(1):506. doi: 10.1186/s12903-023-03206-5. PMID 37480004